CLINICAL TRIAL: NCT01605955
Title: Fingertip Pulse Oximeter Clinical Test
Status: Completed | Type: Observational
Sponsor: Andon Health Co., Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: AndonHealth8
Record Dates: First submitted 2012-05-23; First posted 2012-05-25 (Estimated); Last update posted 2012-05-25 (Estimated); Status verified 2012-04

CONDITIONS: SPO2
Keywords: SPO2

STUDY DESIGN:
Time Perspective: Prospective

GROUPS / COHORTS (2):
- Fingertip Pulse Oximeter: SPO2 measurement range: 70%-99%
- CO-oximeter: SaO2 measurement range: 70%-99%

SUMMARY:
The purpose of this study is to validate the SpO2 accuracy of pulse oximeter equipment in comparison to "gold-standard" measurements of blood SaO2 by a CO-oximeter

ELIGIBILITY:
Inclusion Criteria:

* Subjects participate in the study on a voluntary basis
* All subjects should be in good health at the time of the study. Unless specified otherwise in the protocol, the following values could be applied: COHb<3 %, MetHb<2 %, ctHb>10 g/dl;
* Inclusion criteria should serve the purpose of the study

Exclusion Criteria:

* Smokers or individuals exposed to high levels of carbon monoxide that result in elevated carboxyhaemoglobin levels, unless specific dyshaemoglobins are called for in the study protocol.
* Individuals subject to conditions that result in elevated levels of methaemoglobin, unless specific dyshaemoglobins are called for in the study protocol.
* Subjects who would be placed at undue medical risk associated with any procedures called for in the protocol (e.g. arterial cannulation or hypoxia).
* Age: young person and that of more than 50 years old.

Ages: 25 Years to 32 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: healthy volunteers who consent to induced hypoxia and arterial blood sampling as part of the experimental procedure
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2011-11; Study Completion 2011-12 (Actual)